CLINICAL TRIAL: NCT01722890
Title: CharactHer: A Study of the Molecular and Cytogenetic Characteristics of HER2-positive Breast Cancers to Predict Durable Complete Response After Chemotherapy and Trastuzumab
Brief Title: CharactHer. ICORG 12-09, V3
Status: Terminated | Type: Observational
Why Stopped: As per the HRBs new funding model, HRBs investment will not support costs associated with routine patient care or translational studies, biobanks, patient registries and questionnaires. Therefore, a decision was made to cease further study follow up.
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 12-09
Record Dates: First submitted 2012-10-25; First posted 2012-11-07 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer; TNM Stage II-IV Breast Cancer
Keywords: HER2-positive breast cancer; durable complete response; cytogenetic characteristics; molecular characteristics; trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cohort 1: TNM stage II-IV breast cancer patients with highly trastuzumab-sensitive tumours.
- Cohort 2(Control Group): TNM stage II-IV breast cancer patients with trastuzumab-refractory disease.

SUMMARY:
Primary Objective:

The primary aim of the study is:

1.To identify and validate a panel of molecular and cytogenetic biomarkers able to predict Durable Complete Response (DCR) after chemotherapy and trastuzumab in patients with HER2-positive locally advanced or metastatic breast cancer.

Secondary Objective:

The secondary aims of the study are:

1. To perform a comprehensive exploration of the molecular and cytogenetic characteristics of DCR patients to identify any possible correlation between the tumour's biological and cytogenetic characteristics and the degree of clinical response to trastuzumab;
2. To produce data in preparation for further translational studies on HER2-positive breast cancer.

DETAILED DESCRIPTION:
Type of Study: Translational

This is a pilot retrospective laboratory-based cohort study.

Eligible patients will be identified at each one of the participating institutions by a systematic cross-matching of the datasets of Medical Oncology, Pathology and Pharmacy Departments.

Patient Population:

Cohort 1: TNM stage II-IV breast cancer patients with highly trastuzumab-sensitive tumours.

Cohort 2: (Control group) TNM stage II-IV breast cancer patients with trastuzumab-refractory disease.

ELIGIBILITY:
Inclusion criteria for Cohort 1:

1. Histologically proven AJCC TNM stage II-IV invasive breast cancer
2. HER2-positivity defined as score 3+ on IHC and/or with HER2/neu amplification on FISH test (HER2/CEP17 ratio >2.0 on PathVysion test)
3. Evidence of complete response (CR) according to RECIST 1.1 criteria lasting for at least 36 months (for stage IV patients only) following a first-line chemotherapy and trastuzumab
4. Pathological Complete Response (pCR) following a neo-adjuvant chemotherapy (CT) and trastuzumab (for stage II-III patients only). pCR is defined as no evidence of residual invasive carcinoma in the breast (ductal carcinoma in situ (DCIS) is allowed) AND in all the examined lymph nodes (micro-metastases and isolated tumour cells are not allowed).
5. At least one FFPE archived tissue sample from the primary tumour and/or a metastatic site(s) available for laboratory analyses
6. Adequate follow up information

Inclusion criteria for Cohort 2:

1. Histologically proven AJCC TNM stage II-IV invasive breast cancer
2. HER2-positivity defined as score 3+ on IHC and/or with HER2/neu amplification on FISH test (HER2/CEP17 ratio>2.0 on PathVysion test)
3. Progression of disease according to RECIST 1.1 while receiving trastuzumab (in association with chemotherapy or as single agent as maintenance therapy) or within 6 months from last dose of trastuzumab (for stage IV patients only)
4. Residual invasive tumour in the breast larger than 2cm and /or at least one micro- or macro-metastasis in the axillary lymph nodes following pre-operative trastuzumab-containing chemotherapy (for stage II-III patients only)
5. At least one FFPE archived tissue sample from the primary tumour and/or a metastatic site(s) available for laboratory analyses
6. Adequate follow up information

Exclusion Criteria:

1. Any deviation from the above mentioned Inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of two separate cohorts of patients with HER2-positive breast cancer that will be analysed based on their responsiveness to trastuzumab-containing chemotherapy. Cohort 1 will include patients with TNM stage II-IV breast cancer with highly trastuzumab-sensitive tumours. Results of laboratory analyses from Cohort 1 will be matched with those from Cohort 2 (Control group) that includes patients at the same TNM clinical stages but with trastuzumab-refractory disease.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Panel of molecular and cytogenetic biomarkers able to predict Durable Complete Response (DCR) after chemotherapy and trastuzumab in patients with HER2-positive locally advanced or metastatic breast cancer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Gullo, Medicine and Surgery, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (2):
- St. Vincents University Hospital, Dublin, Ireland
- Humanitas Cancer Centre Milan, Milan, Italy

REFERENCES:
- [Derived] Walsh N, Andrieu C, O'Donovan P, Quinn C, Maguire A, Furney SJ, Gullo G, Crown J. Whole-exome sequencing of long-term, never relapse exceptional responders of trastuzumab-treated HER2+ metastatic breast cancer. Br J Cancer. 2020 Oct;123(8):1219-1222. doi: 10.1038/s41416-020-0999-z. Epub 2020 Jul 27. PMID 32713940